CLINICAL TRIAL: NCT01175941
Title: A Double-blind, Randomized, Placebo-controlled, Cross Over Study in Patient Volunteers With Faecal Incontinence to Evaluate the Effect on Rectal Compliance, Rectal Sensitivity, Recto-anal Inhibitory Reflex, Sphincter Pressures, Safety and Tolerability of a Daily Rectal Application of a 10 mg NRL001 Suppository for Seven Consecutive Days
Brief Title: Effect of 7 Days of Dosing With a 10 mg Rectal Suppository of NRL001in Patients With Faecal Incontinence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NRL001-01/2010 (MANO)
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NRL001 (Experimental): 10 mg NRL001 in a 2 g suppository
  Interventions: Drug: NRL001
- Placebo (Placebo Comparator): Matched placebo control
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: NRL001 — 10 mg NRL001 in a 2 g suppository, administered once daily for 7 days
  Arms: NRL001
Drug: Placebo control — Matched placebo - administered as a 2 g suppository, once daily for 7 days
  Arms: Placebo

SUMMARY:
This is a study to examine the effect of alpha adrenergic stimulation of the anal canal and rectum on parameters affecting the control of defecation in subjects with faecal incontinence. The study will investigate the effects of rectal suppositories containing 10 mg NRL001 given for seven days, once daily. Rectal compliance and median anal resting pressure will be considered the primary objective of the study. A pharmacokinetic evaluation plus safety and tolerability assessment including monitoring of electrocardiograms (ECGs), blood pressure and heart rate will also be evaluated as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient volunteers aged 40 to 85 years without clinically significant or uncontrolled cardiovascular, renal or hepatic disease (as determined by medical history, physical examination, laboratory test values, vital signs, and electrocardiograms [ECGs] at screening)
* Patients with mild/moderate passive faecal incontinence based on clinical symptomology and demonstrating the following criteria:
* ARP ≥20mmHg and ≤80mmHg
* Intact IAS as demonstrated by endoanal ultrasound
* Rectal capacity ≥150ml
* Cleveland Clinic Score ≥6 and ≤ 15
* Body mass index (BMI) ≥ 16 and ≤ 32
* Able and willing to receive rectal treatments
* Able to voluntarily provide written informed consent to participate in the study
* Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol
* Female volunteers must be either postmenopausal (for at least one year and confirmed by serum FSH at screening), or surgically sterile, practising true sexual abstinence, or using Investigator-approved methods of contraception throughout the study until after post study physical examination and have a negative pregnancy test at screening
* Must be willing to consent to have data entered into The Over-Volunteering Prevention System

Exclusion Criteria:

* Patients with FI related to anatomical and/or traumatic sphincter defects
* Presence of any significant or uncontrolled cardiovascular, pulmonary, hepatic, renal, immunologic, neurological or psychiatric disease
* Concomitant ano-rectal conditions or diseases assessed as potentially interfering with the study medication by the Investigator (e.g. concomitant haemorrhoids, anal fissures). Conditions considered not interfering with the study medication are allowed
* Clinically relevant ECG-abnormalities with evident QTc prolongation and/or acute arrhythmia
* Current or history of drug or alcohol abuse
* Use of any disallowed concomitant medication, including over-the-counter items within 30 days prior to study drug administration until the end of the study
* Use of any medication in the last 30 days applied via the rectum
* Use of any medication currently or within the last 30 days which the investigator believes may affect the study participation or results
* Unstable regimen of any statin, hypertensive or diuretic medication (patient volunteers must be on a stable regimen for at least 2 months)
* Participation in a clinical drug study during the 90 days preceding the initial dose in this study
* History of any allergy to nifedipine or any alpha-adrenoceptor antagonist or latex
* Consumption of alcoholic beverages within 24 hours prior to each dosing
* Patient volunteers who are considered not competent to consent to the trial or score less than 25 on the MMSE®
* Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mean anal resting pressure and rectal compliance | 7 days

SECONDARY OUTCOMES:
Rectal sensitivity | 7 days
Adverse events | 7 days
Plasma concentration over time | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Simpson, MD, Principal Investigator — Nottingham University Hospital
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom